CLINICAL TRIAL: NCT01165502
Title: Single-centre, Randomised, Double-blind, Placebo-controlled Clinical Study to Investigate Safety and Tolerability and Pharmacokinetics of Multiple Ascending Doses of CM3.1-AC100 in Healthy Male Volunteers
Brief Title: Clinical Study to Investigate Safety and Tolerability and Pharmacokinetics of Multiple Ascending Doses of CM3.1-AC100 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CellMed AG, a subsidiary of BTG plc. (Industry)
Responsible Party: Dr. Peter Geigle, CellMed AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CellMed CM3.1-AC100/02; 2010-020512-11 (EudraCT Number)
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: MAD study CM3.1-AC100; Healthy men, age 18 - 50

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CM3.1-AC100 (Experimental): Compound CM3.1-AC100 s.c.
  Interventions: Drug: CM3.1-AC100
- Placebo (Placebo Comparator): Placebo for compound CM3.1-AC100 s.c.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CM3.1-AC100 — MAD study with repeated subcutaneous (sc) doses
  Arms: CM3.1-AC100
Drug: Placebo — Placebo for compound CM3.1-AC100 s.c.
  Arms: Placebo

SUMMARY:
The primary objective is to assess the safety and tolerability of the GLP-1 peptide analogue CM3.1-AC100 after repeated subcutaneous (sc) doses.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent prior to any study specific procedures;
* Male volunteer aged 18 to 50 years at Screening, both inclusive;
* Body weight between 60.0 to 100.0 kg (both inclusive) and BMI 19 to 29.9 kg/m2 (both inclusive)

Exclusion Criteria:

* Any history or presence of a clinically relevant disease as judged to be relevant by the Investigator: cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, haematological, neurologic, psychiatric, systemic, ocular or infectious disease and any acute infectious disease or signs of acute illness;
* Blood donation within 3 month before administration of the IP;
* Presence or history of drug allergy, or allergic disease diagnosed and treated by a physician

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety measurements (Adverse events, ECG recordings, blood pressure, pulse, body temperature, laboratory variables, local tolerability, Nausea Intensity, anti- CM3.1-AC100 antibodies) | Safety will be monitored continously and safety assessments will be made on several occasions throughout the whole study

SECONDARY OUTCOMES:
Pharmacokinetic samples for CM3.1-AC100 | Intense PK-sampling during the 15 hours following administration of CM3.1-AC100 during day 1 and day 7
  Pharmacokinetics:
  Following the first dosing on Day 1:
  AUC, AUC0-t, AUC0-9h, Cmax, tmax, t1/2λz, λz, CL/F, Vz/F of CM3.1-AC100.
  Following multiple dosing on Day 7:
  AUCss, AUCss,0-t, AUCss,0-9h, Css,max, Css, min, tss,max, t1/2λz,ss, λz,ss, CLss/F, Vz,ss/F, of CM3.1-AC100.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Geigle, Dr. med., Study Chair — CellMed AG, a subsidiary of BTG plc.
Locations (1):
- Parexel International GmbH, Berlin, State of Berlin, Germany